CLINICAL TRIAL: NCT06028321
Title: Two Part Study to Assess Comparative Bioavailability, Pharmacokinetics of a Single Dose of ACM-001.1, Two Single Doses of Pindolol (Part1) Followed by Evaluation of Steady State Pharmacokinetics, Pharmacodynamics of ACM-001.1 in HV (Part2)
Brief Title: Study of Comparative Bioavailability and Pharmacokinetics of ACM-001.1) and Pindolol in Healthy Volunteers (HV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actimed Therapeutics Ltd (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ACM-2021-1-CT; QSC205141 (Other: Quotient Sciences)
Record Dates: First submitted 2023-07-06; First posted 2023-09-08 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Cachexia
MeSH Terms: conditions — Cachexia | interventions — Pindolol

STUDY DESIGN:
Intervention Model Description: Part 1: part - blinded, part randomized, partial cross- over study. Group 1: double - blinded and randomized to two treatment sequences in a two period cross- over.
  Group 2: open label, non-randomized and in parallel with Group 1. Part 2: single-blind (subject blinded), randomized, parallel-group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part 2 was single - blind study (subject blinded). Masking was not triple for all parts of the study or all arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1 Group1 (AB) (Experimental): Part 1 Group1 Subjects were randomised to two treatment regimens (A and B) and received treatment sequence AB in a 2-period cross over.
  Regimen A = 15 mg ACM-001.1 and matching placebo. Regimen B = 30 mg pindolol.
  Interventions: Drug: Part 1 Group 1 Regime A (ACM-001.1); Drug: Part 1 Group 1 Regimen B (Pindolol); Other: Part 1 Group 1 Regimen A (Placebo)
- Part 1 Group 1 (BA) (Experimental): Subjects were randomised to two treatment regimens (A and B) and received treatment sequence BA in a 2-period cross over.
  Regimen B = 30 mg pindolol. Regimen A = 15 mg ACM-001.1 and matching placebo.
  Interventions: Drug: Part 1 Group 1 Regime A (ACM-001.1); Drug: Part 1 Group 1 Regimen B (Pindolol); Other: Part 1 Group 1 Regimen A (Placebo)
- Part 1 Group 2 (C) (Experimental): Subjects were non-randomised; received regimen C in parallel with Group 1 in a single period.
  Regimen C = 15 mg pindolol.
  Interventions: Drug: Part 1 Group 2 Regimen C (Pindolol)
- Part 2 Group D (Experimental): Subjects received one of the four regimens over a four day treatment period. Regimen D = 20 mg pindolol BID (bis in die) for four days.
  Interventions: Drug: Part 2 Group D (Pindolol)
- Part 2 Group E (Experimental): Subjects received one of the four regimens over a four day treatment period. Regimen E = 5 mg ACM-001.1 and placebo BID for four days.
  Interventions: Drug: Part 2 Group E (ACM-001.1); Other: Part 2 Group E (Placebo)
- Part 2 Group F (Experimental): Subjects received one of the four regimens over a four day treatment period. Regimen F = 10 mg ACM-001.1 and placebo BID for four days.
  Interventions: Drug: Part 2 Group F (ACM-001.1 ); Other: Part 2 Group F (Placebo)
- Part 2 Group G (Experimental): Subjects received one of the four regimens over a four day treatment period. Regimen G = 15 mg ACM-001.1 and placebo BID for four days.
  Interventions: Drug: Part 2 Group G (ACM-001.1); Other: Part 2 Group G ( Placebo)

INTERVENTIONS:
Drug: Part 1 Group 1 Regime A (ACM-001.1) — Drug: ACM-001.1 immediate release tablets for oral use and matching placebo, and pindolol tablets for oral use.
  Subjects randomised to Regimen A received placebo tablets to match the tablet number received by subjects in Regimen B.
  Arms: Part 1 Group 1 (BA); Part 1 Group1 (AB)
Drug: Part 1 Group 2 Regimen C (Pindolol) — Drug: Pindolol tablets for oral use.
  Arms: Part 1 Group 2 (C)
Drug: Part 2 Group D (Pindolol) — Drug: Pindolol tablets for oral use. Subjects were dosed over a four day treatment period twice daily. Subjects receiving ACM-001.1 in regimens E, F and G also received placebo tablets to match the tablet number received by subjects receiving pindolol in Regimen D.
  Arms: Part 2 Group D
Drug: Part 2 Group E (ACM-001.1) — Drug: ACM-001.1 immediate release tablets for oral use and matching placebo. Subjects were dosed over a four day treatment period twice daily. Subjects receiving ACM-001.1 in regimens E, F and G also received placebo tablets to match the tablet number received by subjects receiving pindolol in Regimen D.
  Arms: Part 2 Group E
Drug: Part 2 Group F (ACM-001.1 ) — Drug: ACM-001.1 immediate release tablets for oral use and matching placebo. Subjects were dosed over a four day treatment period twice daily. Subjects receiving ACM-001.1 in regimens E, F and G also received placebo tablets to match the tablet number received by subjects receiving pindolol in Regimen D.
  Arms: Part 2 Group F
Drug: Part 2 Group G (ACM-001.1) — Drug: ACM-001.1 immediate release tablets for oral use and matching placebo. Subjects were dosed over a four day treatment period twice daily. Subjects receiving ACM-001.1 in regimens E, F and G also received placebo tablets to match the tablet number received by subjects receiving pindolol in Regimen D.
  Arms: Part 2 Group G
Drug: Part 1 Group 1 Regimen B (Pindolol) — Drug: pindolol tablets for oral use. Subjects randomised to Regimen A received placebo tablets to match the tablet number received by subjects in Regimen B.
  Arms: Part 1 Group 1 (BA); Part 1 Group1 (AB)
Other: Part 1 Group 1 Regimen A (Placebo) — Placebo for oral use. Subjects randomised to Regimen A received placebo tablets to match the tablet number received by subjects in Regimen B.
  Arms: Part 1 Group 1 (BA); Part 1 Group1 (AB)
Other: Part 2 Group E (Placebo) — Placebo for oral use. Subjects were dosed over a four day treatment period twice daily.
  Subjects receiving ACM-001.1 in regimens E, F and G also received placebo tablets to match the tablet number received by subjects receiving pindolol in Regimen D.
  Arms: Part 2 Group E
Other: Part 2 Group F (Placebo) — Placebo for oral use. Subjects were dosed over a four day treatment period twice daily. Subjects receiving ACM-001.1 in regimens E, F and G also received placebo tablets to match the tablet number received by subjects receiving pindolol in Regimen D.
  Arms: Part 2 Group F
Other: Part 2 Group G ( Placebo) — Placebo for oral use. Subjects were dosed over a four day treatment period twice daily. Subjects receiving ACM-001.1 in regimens E, F and G also received placebo tablets to match the tablet number received by subjects receiving pindolol in Regimen D.
  Arms: Part 2 Group G

SUMMARY:
The aim of this early phase two-part study was to compare the bioavailability (BA) pharmacokinetics (PK) and pharmacodynamics (PD) of racemic pindolol with the benzoate salt of the S-enantiomer of pindolol (ACM-001.1) and provide safety information. A total of 51 healthy male and female subjects were enrolled, and 48 healthy subjects completed the study.

Part 1 consisted of two Groups to compare BA and PK, Group 1 received two treatment sequences of a single dose of ACM-001.1 versus racemic pindolol; Group 2 ran in parallel with Group 1 and assessed the PK of a single dose of racemic pindolol in a single period.

Part 2 consisted of four groups, to evaluate the steady state PK and PD of ACM-001.1 with multiple ascending doses over 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females
* Aged 20 to 45 years inclusive at the time of signing informed consent
* Body Mass Index (BMI) of 18.0 to 30.0 kg/m2 as measured at screening
* Weight of 50 to 100 kg at screening

Exclusion Criteria:

* Subjects who had received any investigational medicinal product in a clinical research study within the 90 days prior to Day 1,
* Subjects for whom pindolol was contraindicated: hypersensitivity to the active substance or to any of its listed excipients.
* Evidence of current Severe Acute Respiratory Coronavirus 2 infection.
* History of any drug or alcohol abuse in the past 2 years.
* Females of childbearing potential who were pregnant or lactating.
* History of clinically significant cardiovascular disease, Raynaud's disease or phenomenon, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder.
* Subjects who were found to have mean heart rate less than 50 bpm at rest or mean systolic blood pressure (BP) less than 100 mmHg or mean diastolic heart rate less than 50 mmHg.
* Subjects who were taking, or had taken, any prescribed or over-the-counter drug or herbal remedies (other than paracetamol, hormonal replacement therapy/hormonal contraception). Pindolol should not be taken in conjunction with agents which inhibit calcium transport.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Part 1 Composite of PK parameters following single doses | Up to 5 days
  Comparative bioavailability of S- pindolol and pindolol include: area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinite].
Part 1 PK parameters following single doses | Up to 5 days
  Comparative bioavailability of S- pindolol and pindolol include:maximum observed concentration (Cmax)
Part 1 PK parameters following single doses | Up to 5 days
  Comparative bioavailability of S- pindolol and pindolol include:time of occurrence of Cmax (Tmax)
PK parameters following single doses | Up to 5 days
  Comparative PK parameters of S- pindolol and racemic pindolol include: area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinite]).
PK parameters following single doses | Up to 5 days
  Comparative PK parameters of S- pindolol and racemic pindolol include: maximum observed concentration (Cmax)
PK parameters following single doses | Up to 5 days
  Comparative PK parameters of S- pindolol and racemic pindolol include: t time of occurrence of Cmax (Tmax)
Stoichiometric dose relationship measured using PK parameters following single doses | Up to 5 days
  PK parameters of S- pindolol and racemic pindolol include: area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinite])
Stoichiometric dose relationship measured using PK parameters following single doses | Up to 5 days
  PK parameters of S- pindolol and racemic pindolol include: maximum observed concentration (Cmax).
Part 2 Composite of PK parameters following multiple doses in plasma | Up to 6 days
  PK parameters of S- pindolol/racemic pindolol:Area under the curve for interval between doses (tau) (AUC(0 tau);Area under the concentration-time curve from time zero (pre-dose) to last time of measurable concentration (AUC[0-t])
Part 2 Composite of PK parameters following multiple doses in plasma | Up to 6 days
  PK parameters of S- pindolol/racemic pindolol: Maximum observed concentration (Cmax),
Part 2 Composite of PK parameters following multiple doses in plasma | Up to 6 days
  PK parameters of S- pindolol/racemic pindolol: Time to first occurrence of Cmax from plasma concentration-time data(Tmax).
Pharmacodynamics of ACM-001.1: Cardiovascular vital parameter- heart rate | Up to 6 days
  Heart rate (beats per minute)
Cardiovascular vital parameter- blood pressure | Up to 6 days
  Systolic blood pressure (mmHG) and diastolic blood pressure (mmHG)
Serum biomarker- DHEA/Cortisol | Day 1 at pre-dose. Day 4 at pre-dose, 1.5 hours
  Dehydroepiandrosterone (DHEA)/Cortisol (ng/mL). Serum concentrations were determined using validated analytical method.
Serum biomarker- Myostatin | Day 1 at pre-dose. Day 4 at pre-dose, 1.5 hours.
  Myostatin (pg/mL).Serum concentrations were determined using validated analytical method.
Serum biomarker- Folistatin | Day 1 at pre-dose. Day 4 at pre-dose, 1.5 hours.
  Folistatin (pg/mL).Serum concentrations were determined using validated analytical method.
Serum biomarker-IGF1 | Day 1 at pre-dose. Day 4 at pre-dose, 1.5 hours.
  Insulin-like growth factor (IGF)1 (pg/mL).Serum concentrations were determined using validated analytical method.
Serum biomarker - (Type 3 procollagen peptide) PIIINP | Day 1 at pre-dose. Day 4 at pre-dose, 1.5 hours.
  PIIINP (pg/mL).Serum concentrations were determined using validated analytical method.
Serum biomarker - monokine-induced by gamma interferon (MIG/CXL9) Leptin | Day 1 at pre-dose. Day 4 at pre-dose, 1.5 hours.
  Leptin (pg/mL).Serum concentrations were determined using validated analytical method.
Serum biomarker - epithelial neutrophil activating peptide 78 (ENA78) | Day 1 at pre-dose. Day 4 at pre-dose, 1.5 hours.
  ENA78 (pg/mL).Serum concentrations were determined using validated analytical method.
Serum biomarker - Ghrelin | Day 1 at pre-dose. Day 4 at pre-dose, 1.5 hours.
  Ghrelin (pg/mL).Serum concentrations were determined using validated analytical method.
Serum biomarker - Growth Hormone Receptor Hormone | Day 1 at pre-dose. Day 4 at pre-dose, 1.5 hours.
  Growth Hormone Receptor Hormone (ng/mL).Serum concentrations were determined using validated analytical method.
Serum biomarker - Somatostatin | Day 1 at pre-dose (baseline). Day 4 at pre-dose, 1.5 hours.
  Somatostatin (pg/mL).Serum concentrations were determined using validated analytical method.

SECONDARY OUTCOMES:
Part 1 Composite PK parameters in urine following single doses | Up to 5 days
  PK parameters of S-pindolol, R-pindolol and pindolol: Amount excreted (Ae), Cumulative amount excreted (CumAe), Fraction of dose excreted (%Ae) and Cumulative fraction of dose excreted (%CumAe)
Part 2 Composite PK parameters in urine following multiple doses and pindolol | Up to 7 days
  PK parameters of S-pindolol, R-pindolol and pindolol: Amount excreted (Ae), Cumulative amount excreted (CumAe), Fraction of dose excreted (%Ae) and Cumulative fraction of dose excreted (%CumAe)
Part 1 and Part 2 Analysis of S-pindolol and R-pindolol concentrations in plasma for any in vivo conversion | Up to 4 days
  Plasma concentrations were determined using validated analytical methods.
Part 1 Number of participants with adverse events following single doses as a measure of safety and tolerability | From screening: day -28 to follow up call on day 8 (part 1), up to 36 days.
  AEs will be collected from provision of written informed consent until discharge at the follow-up contact.
Part 2 Number of participants with adverse events following single doses as a measure of safety and tolerability | From screening: day -28 to follow up call on day 11 (part 2), up to 39 days.
  AEs will be collected from provision of written informed consent until discharge at the follow-up contact
Part 2 only - Pulmonary function test | Up to 32 days
  Forced expiratory spirometry to determine parameters FEV1, FVC, FEV1/FVC

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences Ltd, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: No